CLINICAL TRIAL: NCT06274021
Title: Shared and Distinct Antispastic Effects of Electrical and Pharmacological Neuromodulation
Brief Title: Neuromodulation to Reduce Muscle Stiffness Following Spinal Cord Injury
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Collaborators: Methodist Rehabilitation Center (Other); The Craig H. Neilsen Foundation (Other)
Responsible Party: Principal Investigator, Matthias J. Krenn, PhD, Assistant Professor, University of Mississippi Medical Center
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: UMMC-IRB-2023-125
Record Dates: First submitted 2023-11-17; First posted 2024-02-23 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Spinal Cord Injuries; Spinal Cord Injury; Spinal Cord Injury Cervical; Spinal Cord Injury Thoracic
Keywords: Spinal Cord Injury; Neuromodulation; Electrical Stimulation; Spinal Cord Stimulation; Spasticity; Transcutaneous Spinal Stimulation; Lower extremity; Transcutaneous spinal cord stimulation; Paralysis; Spinal reflex
MeSH Terms: conditions — Spinal Cord Injuries; Muscle Spasticity; Paralysis | interventions — Baclofen; tizanidine

STUDY DESIGN:
Intervention Model Description: This study employs a crossover design, wherein each participant is systematically administered a sequence of five distinct interventions randomly. This approach ensures that every participant receives each intervention in a unique sequence. The design facilitates within-subject comparisons by minimizing inter-individual variability, as each participant effectively serves as their own control across the study phases. The random assignment of intervention sequences aims to balance potential carryover effects and period effects.
Masking Description: The participants and assessors are kept unaware of which intervention is being administered. For this, the study drugs are designed to be visually identical for all participants, and the intervention and sham stimulation configuration is set without the assessor being present in the room.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transcutaneous spinal stimulation in combination of baclofen/tizanidine/placebo (Experimental): Each participant will receive five distinct interventions:
  * Transcutaneous spinal stimulation at 100 Hz for 30 minutes with a placebo
  * Transcutaneous spinal stimulation at 50 Hz for 30 minutes with a placebo
  * Transcutaneous spinal stimulation at 50 Hz for 30 minutes with a single-dose baclofen
  * Transcutaneous spinal stimulation at 50 Hz for 30 minutes with a single-dose tizanidine
  * Transcutaneous spinal stimulation (sham) for 30 minutes with a placebo
  Interventions: Device: Transcutaneous spinal stimulation at 100 Hz; Device: Transcutaneous spinal stimulation at 50 Hz; Combination Product: Transcutaneous spinal stimulation at 50 Hz and single dose of baclofen; Combination Product: Transcutaneous spinal stimulation at 50 Hz and single dose of tizanidine; Device: Sham transcutaneous spinal stimulation

INTERVENTIONS:
Device: Transcutaneous spinal stimulation at 100 Hz — Transcutaneous spinal stimulation (TSS) is a non-invasive neuromodulation method that uses electrical currents to stimulate sensory fibers. The procedure involves placing surface electrodes midline on the lower back (T11-12 spinal processes) and on each side of the belly button. The stimulation frequency during the intervention is 100 Hz, performed at a sub-motor threshold for 30 minutes.
Device: Transcutaneous spinal stimulation at 50 Hz — Transcutaneous spinal stimulation (TSS) is a non-invasive neuromodulation method that uses electrical currents to stimulate sensory fibers. The procedure involves placing surface electrodes midline on the lower back (T11-12 spinal processes) and on each side of the belly button. The stimulation frequency during the intervention is 50 Hz, performed at a sub-motor threshold for 30 minutes.
Combination Product: Transcutaneous spinal stimulation at 50 Hz and single dose of baclofen — Transcutaneous spinal stimulation (TSS) is a non-invasive neuromodulation method that uses electrical currents to stimulate sensory fibers. The procedure involves placing surface electrodes midline on the lower back (T11-12 spinal processes) and on each side of the belly button. The stimulation frequency during the intervention is 50 Hz, performed at a sub-motor threshold for 30 minutes.
  Study participants will receive a single dose of baclofen, a centrally-acting muscle relaxant belonging to the class of gamma-aminobutyric acid (GABA) analogs. Its primary mechanism involves acting on the GABA receptors in the brain and spinal cord to decrease spasticity. Participants will receive baclofen orally at a single dose of 10 mg.
Combination Product: Transcutaneous spinal stimulation at 50 Hz and single dose of tizanidine — Transcutaneous spinal stimulation (TSS) is a non-invasive neuromodulation method that uses electrical currents to stimulate sensory fibers. The procedure involves placing surface electrodes midline on the lower back (T11-12 spinal processes) and on each side of the belly button. The stimulation frequency during the intervention is 50 Hz, performed at a sub-motor threshold for 30 minutes.
  Study participants will receive a medication called tizanidine, which is an alpha-2 adrenergic agonist. This medication works by inhibiting presynaptic motor neurons, resulting in a reduction of muscle spasticity. It is commonly used to manage spasticity caused by neurological disorders. Each participant will be given a single oral dose of 4 mg of tizanidine as part of this trial.
Device: Sham transcutaneous spinal stimulation — Sham Transcutaneous spinal stimulation (TSS) involves placing two surface electrodes midline on the lower back (T11-12 spinal processes). The stimulation frequency during the intervention is 50 Hz, performed for 30 minutes.

SUMMARY:
People with spinal cord injuries may experience muscle tightness or uncontrollable spasms. This study is being conducted to investigate whether transcutaneous spinal stimulation can improve these symptoms. Transcutaneous spinal stimulation is a non-surgical intervention by applying electrical currents using skin electrodes over the lower back and belly.

The investigators want to see how well the intervention of transcutaneous spinal stimulation performs by testing different levels of stimulation pulse rates. Also, transcutaneous spinal stimulation is compared to muscle relaxants such as baclofen and tizanidine, commonly given to people with spinal cord injuries, to reduce muscle stiffness and spasms. By doing this, the investigators hope to discover if transcutaneous spinal stimulation similarly reduces muscle spasms and stiffness or if combining both methods works best. This could help improve treatment options for people with spinal cord injuries in the future.

DETAILED DESCRIPTION:
The primary questions to be addressed are whether the intervention reduces muscle stiffness and spasms and alters spinal reflexes:

* Using a 100-Hz (a measure of frequency) transcutaneous spinal stimulation is better than using a 50-Hz.
* Transcutaneous spinal stimulation at 50 Hz differs from a single dose of baclofen.
* Transcutaneous spinal stimulation at 50 Hz differs from a single dose of tizanidine.
* Combining the 50 Hz stimulation with either baclofen or tizanidine decreases spasticity more than just taking the medicine alone.

Participants will visit the Methodist Rehabilitation Center in Jackson, Mississippi, six times over a period of 3 to 5 weeks. During the first visit, the overall health and motor and sensory functions will be assessed following a spinal cord injury. For the next five visits, participants will take a study medication (tizanidine, baclofen, or a placebo). After an hour, they will receive a continuous 30-minute transcutaneous spinal stimulation at either 50 Hz, 100 Hz, or sham. The spinal reflexes and clinical assessments will be evaluated before, during, and after each intervention.

ELIGIBILITY:
Inclusion criteria:

* Age 18 years or older
* History of spinal cord injury
* Time since diagnosis longer than six months
* Presence of spasticity in the lower limbs (≥ 3 on the Numerical Rating Scale of Spasticity Severity [range from 0 to 10])
* If needed, agreement to reduce antispastic medication

Exclusion criteria:

* Neurological level of spinal cord injury below T11
* Ventilatory-dependent
* Change in neurological status over the past 2 months
* Rigidity, contraction, or passive range of motion of less than 40 deg in both knee joints
* Botulinum toxin injections in lower extremities in the previous 3 months before enrollment
* Systolic blood pressure at rest lower than 90 mm Hg
* Implanted active devices (e.g., intrathecal baclofen pumps)
* Passive implants (plates, screws) between T11 and L2 vertebras
* Skin conditions precluding placement of electrodes
* Pressure ulcers stage 2 or higher on the gluteal area or lower extremities
* Receiving antibiotics for infections
* Pregnancy
* Difficulty following instructions
* Participation in another study with investigational drugs or devices within the 30 days preceding and during the present study
* Other medical risks/contraindications as determined by the study physicians

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of posterior root reflexes (PRRs) recruitment curves. | Baseline and at post-intervention (100 minutes)
  Change in area under the recruitment curve of PRRs after the intervention compared to the baseline. These reflexes are elicited by transcutaneous spinal stimulation and recorded in key muscles of the lower extremities.
Change from baseline of flexion withdrawal reflex (FWR) response amplitude. | Baseline and at post-intervention (100 minutes)
  Change in the amplitude of the FWR response after the intervention compared to the baseline. The reflex response indicates neural circuitry function and spasticity in individuals with neurological conditions. It is measured by eliciting a motor response through a standardized electrical stimulus and quantifying the change in muscle activity.
Change from baseline of stretch reflex (SR) response amplitude. | Baseline and at post-intervention (100 minutes)
  Change in the amplitude of the SR response after the intervention compared to the baseline. The reflex response indicates spasticity and muscle tone in participants with neurological disorders. The amplitude of the reflex response reflects the muscle's reaction to stretch.
Change from baseline in muscle stiffness as measured by the Modified Ashworth Scale (MAS), | Baseline and at post-intervention (100 minutes)
  Change in cumulative scores of Modified Ashworth Scale in bilaterally five lower extremity muscles (score range: 0 to 40, where higher scores denote worsening outcomes) before and after the 30-minute intervention. The Modified Ashworth Scale is a clinically validated tool that measures resistance during passive soft-tissue stretching and indicates spasticity.
Change from baseline in spasms as measured by the Spinal Cord Assessment Tool for Spastic Reflexes (SCATS). | Baseline and at post-intervention (100 minutes)
  Change in the cumulative score of the Spinal Cord Assessment Tool for Spastic Reflexes, encompassing clonus, flexor spasms, and extensor spasms bilaterally, with a scoring range from 0 to 18, where higher scores denote worsening outcomes. The Spinal Cord Assessment Tool for Spastic Reflexes is a clinical tool designed to evaluate spastic reflexes in individuals with spinal cord injury specifically. It quantitatively measures the severity and pattern of spasticity by assessing involuntary muscle contractions in response to external stimuli.

SECONDARY OUTCOMES:
Change from baseline of posterior root reflexes (PRRs) recruitment curves. | Baseline and at during transcutaneous spinal stimulation (80 minutes)
  Change in area under the recruitment curve of PRRs during transcutaneous spinal stimulation compared to the baseline. These reflexes are elicited by transcutaneous spinal stimulation and recorded in key muscles of the lower extremities.
Change from baseline of flexion withdrawal reflex (FWR) response amplitude. | Baseline and at during transcutaneous spinal stimulation (80 minutes)
  Change in the amplitude of the FWR response during transcutaneous spinal stimulation compared to the baseline. The reflex response indicates neural circuitry function and spasticity in individuals with neurological conditions. It is measured by eliciting a motor response through a standardized electrical stimulus and quantifying the change in muscle activity.
Change from baseline of stretch reflex (SR) response amplitude. | Baseline and at during transcutaneous spinal stimulation (80 minutes)
  Change in the amplitude of the SR response during transcutaneous spinal stimulation compared to the baseline. The reflex response indicates spasticity and muscle tone in participants with neurological disorders. The amplitude of the reflex response reflects the muscle's reaction to stretch.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias J Krenn, Ph.D., Principal Investigator — University of Mississippi Medical Center
Locations (2):
- United States (2):
  - Methodist Rehabilitation Center, Jackson, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi

IPD SHARING:
Plan to Share IPD: No